CLINICAL TRIAL: NCT06571526
Title: Investigating Visual Search Strategies and the Role of Attentional Focus During Psychomotor Gait Re-education in Older Adults at Risk of Falling: Implication for Fall Rehabilitation
Brief Title: External Focus Strategy on Visuomotor Control in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20210525002
Record Dates: First submitted 2024-08-21; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Gait; Fall Risk; Older Adults
Keywords: attentional focus; gait; older adults; visual search

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXT (Experimental)
  Interventions: Behavioral: External focus
- CON (Active Comparator)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: External focus — The training phase consisted of 20 consecutive training trials, with a rest interval of at least 30 seconds between trials. All participants had to circumvent an obstacle during each trial on the 8-m level-ground walkway. During each trial, the general instruction was to focus on a random series of digits ranging from 0 to 9 displayed on monitors placed at the immediate and future destinations of the walkway. Each number was displayed for at least 2 seconds to allow participants to have sufficient time to read them.
  Arms: EXT
Behavioral: Control — The training phase consisted of 20 consecutive training trials, with a rest interval of at least 30 seconds between trials. All participants had to circumvent an obstacle during each trial on the 8-m level-ground walkway. During each trial, the general instruction was to walk to the end of the walkway at your natural pace.
  Arms: CON

SUMMARY:
Only a few studies have adopted external focus strategy as an intervention to mitigate the negative effects of heightened conscious movement processing in older adults. The goal was to investigate whether a single-session intervention (SSI) using external focus strategy could improve gait stability and visual search behaviors during adaptive locomotion among the older population.

Participants were randomly allocated to either an external focus (EXT) or a control group (CON). All participants performed an obstacle circumvention walking task along an 8-m walkway for five trials at pre-intervention (T0), post-intervention (T1), and retention (T2). The training phase included 20 walking trials. EXT focused on digits displayed on monitors at their path destinations, while CON walked naturally without any manipulation.

ELIGIBILITY:
Inclusion Criteria:

* aged 65 or above
* were able to walk independently indoors without walking aids

Exclusion Criteria:

* a total score of less than 24 on the Chinese version of the Mini-Mental State Examination
* a static visual acuity poorer than 20/40 vision
* the presence of any untreated cerebral vascular disease, Parkinson's disease, or any other major neurological deficit

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 112 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Gait stability | pre-test, post-test (the same day, immediately after the single-session intervention), 1 week after post-test (retention)
  Measured by a 3-D motion-capture system. Indicated by the variabilities of temporal and spatial gait parameters
Visual search behavior | pre-test, post-test (the same day, immediately after the single-session intervention), 1 week after post-test (retention)
  Measured by eye tracker.
  Indicated by:
  number of fixation (%) on ground number of fixation (%) on destination number of fixation (%) on obstacle number of fixation (%) on random areas fixation duration (%) on ground fixation duration (%) on destination fixation duration (%) on obstacle fixation duration (%) on random areas

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong